CLINICAL TRIAL: NCT01930383
Title: Circulating Tumor Cells (CTCs) as Biomarkers of Prognosis and Predictors of Efficacy of Drug Therapy for Patients With Hepatocellular Carcinoma
Brief Title: Circulating Tumor Cells for Hepatocellular Carcinoma
Acronym: CTCs for HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201306057RIND; ctcs201305 (Other: Research Ethics Committee)
Record Dates: First submitted 2013-08-20; First posted 2013-08-28 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Carcinoma, Hepatocellular; Neoplasm Circulating Cells
Keywords: biomarkers
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood samples will be separated to blood cells and plasma. Blood cells will be used for isolation and enumeration of CTCs. Plasma will be used to extract DNA to measure molecular aberration (gene mutations related to hepatocarcinogenesis or response of HCC cells to molecular targeted therapy).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Arm A: HCC patients who receive curative surgery or radiofrequency ablation therapy
- Arm B: patients who receive trans-arterial chemoembolization
- Arm C: patients who receive systemic therapy

SUMMARY:
To explore the clinical value of circulating tumor cells (CTCs) measurement for Hepatocellular carcinoma (HCC) patients.

DETAILED DESCRIPTION:
Background:The lack of tumor tissue for drug target and biomarker studies significantly limit the development of novel treatment for advanced HCC. In recent years, circulating tumor cells (CTCs) have been shown to be important prognostic biomarkers of overall survival for patients with breast, prostate, and colorectal cancer after anti-cancer therapy.

Methods and Materials:This project plans to enroll 50 HCC patients who receive curative surgery or radiofrequency ablation therapy, 50 patients who receive trans-arterial chemoembolization, and 50 patients who receive systemic therapy at National Taiwan University Hospital in 24 months for CTCs analysis. The eligible patients will receive blood tests before and after anti-cancer therapy. The blood samples will be separated to blood cells and plasma. Blood cells will be used for isolation and enumeration of CTCs. Plasma will be used to extract DNA to measure molecular aberration (gene mutations related to hepatocarcinogenesis or response of HCC cells to molecular targeted therapy)

1. to explore the correlation between CTCs numbers and other clinical characteristics in HCC patients with different stages;
2. to compare the patterns of molecular aberrations between CTC and HCC tumor tissue in HCC patients who have archival tumor tissue available; and
3. to measure the changes of CTCs numbers and molecular aberrations in HCC patients before and after molecular targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be diagnosed with HCC via one of following methods according to present clinical practice:

  1. Diagnosed as HCC by biopsy or cytology
  2. Patients with chronic hepatitis B or other reason induced liver cirrhosis who have diagnosed as HCC based on a typical contrast enhanced CT or MRI profile with malignant lesion [tumor hyper-vascularization].
* Asian male or female subjects >=20 years of age.
* Child-Pugh class A or B liver function..
* HCC patients who will receive anti-cancer therapy, including surgery, radiofrequency ablation therapy, trans-arterial chemoembolization, or systemic therapy (according to current HCC practice guidelines) at National Taiwan University Hospital.
* Signed informed consent.

Exclusion Criteria:

* Other significant organ disease or condition his/her investigator judged that the subject should not participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Numbers of circulating tumor cells | in 24 months
  CTCs are measured by microfluidic disk platform. They are defined as tumor cells that are circulating in the peripheral blood of patients, which are shed from either the primary tumor or its metastases.

SECONDARY OUTCOMES:
Overall survival | 24 months
Clinical characteristics | in 24 months
  The other clinical characteristics was defined as following characteristics:
  1. Sex
  2. Age
  3. Barcelona-Clinic Liver Cancer[BCLC] staging
  4. alpha feto protein[AFP] level
  5. Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Chiun Hsu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan